CLINICAL TRIAL: NCT05620121
Title: ACute Treatment of Incisional Ventral Hernia: an Italian Collaborative Study
Brief Title: ACute Treatment of Incisional Ventral Hernia
Acronym: ACTIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Camillo (Other)
Responsible Party: Principal Investigator, Lorenzo Crepaz, MD, Principal Investigator, Ospedale San Camillo
Other Study IDs: 2022/0006983/P/IFSC
Record Dates: First submitted 2022-11-04; First posted 2022-11-17 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Incisional Hernia
Keywords: Incisional Hernias; Minimally invasive surgery; Mesh; Emergency; Abdominal wall defects
MeSH Terms: conditions — Incisional Hernia; Emergencies | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive IH surgery: Minimally invasive approach to incisional hernias in non-electice settings
  Interventions: Procedure: Surgery for Incisional hernias
- Laparotomic IH surgery: Laparotomic approach to incisional hernias in non-electice settings
  Interventions: Procedure: Surgery for Incisional hernias

INTERVENTIONS:
Procedure: Surgery for Incisional hernias — Laparoscopic and laparoscopic abdominal wall repair for Incisional Hernia with/without prosthetic material in urgent/emergent settings, with/without direct closure of the defect (IPOM and IPOM +).

SUMMARY:
This observational, retrospective study aims to examine surgical outcomes in non-elective surgery for incisional hernia.

The main questions it aims to answer are:

* 30-day morbidity
* short- and long-term surgical outcomes

Data will be retrospectively collected from participating centers and compared. Researchers will compare surgical outcomes of the minimally invasive and laparotomic approaches to see if there are relevant differences in surgical outcomes.

DETAILED DESCRIPTION:
Incisional abdominal hernias are a common challenge for general surgeons, as a possible natural consequence of a considerable amount of abdominal wall trauma for laparotomic, laparoscopic, endoscopic, or robotic accesses.

In Italy, almost 17.000 cases per year of primitive and incisional hernias are diagnosed, leading to a wide necessity for surgical repair of abdominal wall defects, with a subsequent growing interest in the technical and technological aspects of this kind of surgery.

The real complexity of this kind of disease must be sought in various elements: different abdominal sites, different hernias' content, and a surgical approach that must aim to make abdominal wall repair as valid and definitive as possible.

For these reasons, a growing number of surgeons have ventured into abdominal wall surgery, with encouraging results and with techniques reproducible in many departments, expanding the surgical approach in this specific field, and getting a more anatomical and complete understanding of abdominal wall defects.

In the last years, minimally invasive surgery has taken place more and more, due to the evident advantages in terms of surgical outcomes, increasing the technical laparoscopic, endoscopic, and robotic knowledge worldwide.

Under these conditions, with technical and technological development constantly evolving, many centers started and consolidated a valid cure standard for primitive and incisional abdominal hernias with minimally invasive techniques.

The rationale of a minimally invasive approach to abdominal hernias, as for many other surgical fields, resides in consistent advantages in terms of postoperative pain, surgical site infection ratio, minor length of stay, smaller postoperative complications ratio, and therefore, a partial reduction in costs derived from laparoscopic, endoscopic and robotic equipment.

Indication of a minimally invasive approach to incisional hernias derives principally from the evaluation of the surgical outcomes for those patients who could resent of laparotomic approach for surgical defect repair, counteracting intraoperative technical difficulties for surgeons.

From clinical practice and literature reviews, a minimally invasive approach to incisional hernias in non-elective settings appears nowadays still limited to stable patients, without an excessive intestinal dilatation upstream of intestinal incarceration, with a small-sized wall defect, but without a clear preoperative predictor of surgical outcomes.

The ACTIVE studio (ACute Treatment of Incisional Ventral hErnia) aims to analyze and compare surgical outcomes of a non-elective approach to incisional hernias, with a specific focus on short- and long-term results for both laparotomic and laparoscopic techniques.

Further data aims to outline and compare different surgical techniques used, different prosthetic materials, and different pre and postoperative routines in various centers, in relation to defect features.

Aim of the study

Retrospective and multicentric evaluation of Incisional Hernia (IH) urgent treatment, analyzing and comparing the results of those surgical outcomes and the technical and managing features in various centers based on the scientific knowledge available today. The study's principal endpoint compares the short-term morbidity rate between laparoscopic and laparotomic approaches.

Study Population

All consecutive adult patients admitted to the participating surgical departments who underwent urgent/emergent surgery for Incisional Hernia, in the period between 1st January 2018 and 31st December 2021.

Intervention

Laparoscopic abdominal wall repair for Incisional Hernia with/without prosthetic material in urgent/emergent settings, with/without direct closure of the defect (IPOM and IPOM +).

Comparison

Laparotomic abdominal wall repair for Incisional Hernia with/without prosthetic material in urgent/emergent settings.

Study characteristics

Multicentric, retrospective, observational study. The study will include all the consecutive patients who underwent surgical procedures for IH repair in urgent and emergent settings, in the period between January 2018 and December 2021.

Sample Size

The sample size has been calculated starting from literature data disposable (clinical trials, systematic reviews, international and national guidelines), reaching a morbidity rate after surgery for IH that has been used as a starting point for the present study.

We estimated that a minimum of 200 patients per group (minimally invasive vs. open) would yield a power of 0.80 (1-ß) to establish whether minimally invasive technique for IH surgery in urgent/emergent settings impacted in global postoperative morbidity, using a one-sided significance ɑ level of 0.05 (5%).

Indeed, from the current literature data, the morbidity after IH surgery with open surgery can be estimated at around 12%, while data referring to the laparoscopic approach are at around 5%, with a consequent reduction of overall postoperative morbidity of almost 7% using a minimally invasive approach.

The present analysis has been done with an online power sample size calculator (sealedenvelope.com).

Participating centers

The study once approved by the Ethical Committee of Promoting Center has been proposed to SICE and ISHAWS members, beyond clinicians who answered the previously and appositely created online open survey (https://siceitalia.com/survey-laparoceli/).

Study period

The departments involved in the study will have to enter the requested data from 15th September 2022 to 31st January 2023.

Evaluated features

General features (sex, age, BMI, Charlson Score index, ASA score) Patient clinical status upon admission Incisional hernia features Type of eventual defect repair and prosthetic features Postoperative complications (Clavien-Dindo score), length of stay, 30-day mortality, 30-day morbidity Long-term surgical outcomes

Data collection

All epidemiological, clinical, and surgical data will be collected on a CRF (a Microsoft Excel form) that will be sent via email to only one contact person (Local Lead) of each participating center. Once CRF will be properly filled out, will be sent through a pre-supplied link, that only allows the upload of files, to a protected Dropbox account, managed by Delphi International (collaborating with the SICE secretariat). Subsequently, data will be recovered from Principal Investigator, and locally elaborated.

All clinical data inserted will be anonymous.

Funding

This research has not received any specific grant from funding agencies in the public, commercial, or not-for-profit sectors.

Financial and Insurance

Not applicable.

Statistical analysis

In the study results, the dichotomous variables will be expressed as numbers and percentages, while continuous variables will be expressed as mean and SD for normal data distributions, or median and IQR for non-normal data distributions (minimum and maximum values). Student's t-test or ANOVA will be used for inferential statistical analysis of quantitative data.

Binary logistic regression models will be used to investigate clinical attitudes (like the surgical technique), and basic, laboratory, and radiological variables, predictive of morbidity and mortality. A value of P < 0.05 will be considered statistically significant.

Ethical aspects

This is a national observational study; it will not attempt to change or modify the clinical practice of the participating physicians. The study will meet and conform to the standards outlined in the Declaration of Helsinki and Good Epidemiological Practices. Every clinical center attending the study is responsible for Ethics Committee approval depending on the local policy for observational and non-interventional studies. All surgeons involved in the patients' recruitment will be included in the research authorship.

Publication policy

The Local Lead and two Collaborators from each center will be listed as Co-authors in the final publications. Data will be published as a pool from all participating surgical units. Data that emerged from the ACTIVE study will be published irrespective of findings. Results will be published on ClinicalTrials.Gov and each manuscript that is generated based on the registry will be disseminated to all participating centers before final publication.

Data management

Every local investigator is responsible for entering data on an online case report form for every patient included in the study.

Informed consent

Due to its retrospective design, this observational study will not attempt to change or modify the laboratory or clinical practices of the participating physicians. Consequently, informed consent will not be required.

Safety issues

None.

Authors

A maximum of two authors per participating center will be listed as authors in final publications.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes,
* ≥ 18 years old
* IH surgery in urgent/emergent settings
* open or minimally invasive surgical approach

Exclusion Criteria:

* Pregnant women
* ≥ 80 years old patients
* primitive abdominal wall hernias
* perineal or parastomal hernias

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients admitted to the participating surgical departments who underwent urgent/emergent surgery for Incisional Hernia, in the period between 1st January 2018 and 31st December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
30-day morbidity | first 30 days after surgery
  (according to Clavien-Dindo classification) in patients who underwent abdominal wall repair for Incisional Hernia with/without prosthetic material in urgent/emergent settings, with the laparoscopic or the laparotomic approach.

SECONDARY OUTCOMES:
30-day mortality | first 30 days after surgery
  Mortality during the study period
30-day hospital readmission rate | first 30 days after surgery
  hospital readmission within 30-days from discharge, due to surgery-related complications
Reoperation rate | 01 january 2018 - 31 December 2021
  surgical interventions along the study period, due to complications or recurrences of IH surgery
Short-term IH recurrence | 01 january 2018 - 31 December 2021
  Recurrence rate within the first year after surgery
Long-term IH recurrence | 01 january 2018 - 31 December 2021
  Recurrence rate after the first year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Crepaz, Study Director — Ospedale San Camillo
Locations (1):
- Lorenzo Crepaz, Trento, Italy

IPD SHARING:
Plan to Share IPD: No
There is no intention to share data for other reserchers

REFERENCES:
- [Background] Stoppa RE. The treatment of complicated groin and incisional hernias. World J Surg. 1989 Sep-Oct;13(5):545-54. doi: 10.1007/BF01658869. PMID 2683400
- [Background] Ramirez OM, Ruas E, Dellon AL. "Components separation" method for closure of abdominal-wall defects: an anatomic and clinical study. Plast Reconstr Surg. 1990 Sep;86(3):519-26. doi: 10.1097/00006534-199009000-00023. PMID 2143588
- [Background] Hartog FPJD, Sneiders D, Darwish EF, Yurtkap Y, Menon AG, Muysoms FE, Kleinrensink GJ, Bouvy ND, Jeekel J, Lange JF. Favorable Outcomes After Retro-Rectus (Rives-Stoppa) Mesh Repair as Treatment for Noncomplex Ventral Abdominal Wall Hernia, a Systematic Review and Meta-analysis. Ann Surg. 2022 Jul 1;276(1):55-65. doi: 10.1097/SLA.0000000000005422. Epub 2022 Feb 18. PMID 35185120
- [Background] Rosen MJ, Jin J, McGee MF, Williams C, Marks J, Ponsky JL. Laparoscopic component separation in the single-stage treatment of infected abdominal wall prosthetic removal. Hernia. 2007 Oct;11(5):435-40. doi: 10.1007/s10029-007-0255-y. Epub 2007 Jul 24. PMID 17646896
- [Background] Cox TC, Pearl JP, Ritter EM. Rives-Stoppa incisional hernia repair combined with laparoscopic separation of abdominal wall components: a novel approach to complex abdominal wall closure. Hernia. 2010 Dec;14(6):561-7. doi: 10.1007/s10029-010-0704-x. Epub 2010 Jul 27. PMID 20661611
- [Background] Poelman M, Apers J, van den Brand H, Cense H, Consten E, Deelder J, Dwars B, van Geloven N, de Lange E, Lange J, Simmermacher R, Simons M, Sonneveld E, Schreurs H, Bonjer J. The INCH-Trial: a multicentre randomized controlled trial comparing the efficacy of conventional open surgery and laparoscopic surgery for incisional hernia repair. BMC Surg. 2013 Jun 7;13:18. doi: 10.1186/1471-2482-13-18. PMID 24499061
- See also: Trattamento laparoscopico del laparocele ed ernie ventrali - Linee guida italiane, SICE — https://snlg.iss.it/wp-content/uploads/2022/02/LG-478-SICE_laparocele.pdf